CLINICAL TRIAL: NCT07308184
Title: A Multi-center, Randomized, Double-Blind, Placebo Controlled, Parallel, Phase 3 Bridge Study to Evaluate the Efficacy and Safety of IN-B00009 Injection in Patients With T2DM Inadequately Controlled by Diet and Exercise Alone
Brief Title: Bridge Study to Evaluate the Efficacy and Safety of IN-B00009 Injection in Patients With T2DM Inadequately Controlled by Diet and Exercise Alone
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN_ECN_302
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Diabetes (DM); Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-B00009 (Experimental)
  Interventions: Drug: IN-B00009
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IN-B00009 — Test drug
  Arms: IN-B00009
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
This Phase 3 Bridge study is designed to evaluate the efficacy and safety of IN-B00009 Injection in Patients with T2DM Inadequately Controlled by Diet and Exercise Alone

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, Parallel, Phase 3 Bridge study. If the subjects are ultimately determined to meet all inclusion/exclusion criteria based on the results of the pre-randomization testing conducted at Visit 3, they are stratified based on HbA1c (≤ 8.5%, > 8.5%) and randomly assigned to either the study group or the placebo group in a 1:1 ratio at Visit 4. Subjects will receive the investigational product once weekly for up to 24 weeks.

During the 24-week treatment period, the study group will begin with IN-B00009 injection at an initial dose of 0.3 mg and increase the dose at 4-week intervals to reach a target dose of 1.2 mg. After reaching the target dose, the dose will be maintained. The placebo group will receive the same volume of placebo as the study group at each time point.

* Duration of Administration / Study Group / Placebo Group 4 weeks(week 0 ~ week 3) / IN-B00009 inj. 0.3 mg / Placebo 0.15 mL 4 weeks(week 4 ~ week 7) / IN-B00009 inj. 0.6 mg / Placebo 0.3 mL 16 weeks(week 8 ~ week 23) / IN-B00009 inj. 1.2 mg / Placebo 0.6 mL

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 19 to 75 years at the time of written consent
2. Subjects with a BMI ≥ 20 kg/m² and ≤ 35 kg/m² at the screening visit

   ☞BMI (kg/m²) = Weight (kg) / Height (m)²
3. Among subjects who have been diagnosed with T2DM at least 12 weeks ago and have followed a stable diet and exercise program for at least 8 weeks prior to the screening visit, those who meet any of the following criteria:

   * Those who have not administered hypoglycemic agents within the past 12 weeks
   * Those who have administered oral hypoglycemic agents within the past 12 weeks, but have not administered them within 5 weeks prior to the screening visit
4. Subjects with HbA1c levels of 7.5% to 11.0% at the screening visit and 7.0% to 10.5% before randomization
5. Subjects with fasting plasma glucose (FPG) levels ≤ 250 mg/dL (13.9 mmol/L) at the screening visit and pre-randomization testing
6. Subjects who are able to self-monitor blood glucose levels and record subject diary cards during the study
7. Subjects who agree to use medically acceptable contraceptive methods (including those medically incapable of pregnancy) during the study
8. Subjects who are able to understand and follow instructions and participate throughout the study

Exclusion Criteria:

1. Subjects who have been diagnosed with type 1 diabetes mellitus (T1DM) or diabetes due to a genetic defect or exocrine pancreatic dysfunction
2. Subjects who have been administered GLP-1 analogues or DPP-4 inhibitors within 12 weeks prior to the screening visit
3. Subjects who have used insulin within 24 weeks prior to the screening visit (excluding the short-term use for the treatment of hyperglycemia symptoms within a total of 14 days)
4. Subjects with a history of diabetic ketoacidosis, hyperosmolar hyperglycemia, or diabetic lactic acidosis within 24 weeks prior to the screening visit
5. Subjects with a history of severe chronic diabetic complications (proliferative diabetic retinopathy or diabetic maculopathy, diabetic peripheral neuropathy, etc.) within 24 weeks prior to the screening visit
6. Subjects with a history of level 3 severe hypoglycemia within 24 weeks, or two or more events of level 2 hypoglycemia (blood glucose < 54 mg/dL) within 4 weeks prior to the screening visit
7. Subjects with a history of severe trauma, infection, or surgery that may affect glycemic control within 4 weeks prior to the screening visit
8. Subjects with a history of uncontrolled hyperthyroidism or hypothyroidism (However, those with 0.4 uIU/mL ≤ TSH ≤ 6.8 uIU/mL at the screening visit, who have been taking a stable dose of thyroid hormone medication for the past 12 weeks, and whose dose is unlikely to change during the study can participate.)
9. Subjects with a history (including family history) of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2)
10. Subjects who have received medical or non-medical weight management, including weight management medications or products, within 12 weeks prior to the screening visit, or whose weight percent change confirmed by clinical interview exceeded 5%
11. Subjects with at least one of the following medical histories confirmed within 24 weeks prior to the screening visit

    * NYHA class III or IV heart failure
    * Coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI)
    * Ischemic heart disease (acute myocardial infarction, unstable angina, etc.)
    * Severe cerebrovascular disease (cerebral infarction, cerebral hemorrhage, etc.), transient ischemic attack (TIA)
12. Subjects with a history of uncontrolled respiratory disease (chronic obstructive pulmonary disease, bronchial asthma, active tuberculosis, etc.) within 24 weeks prior to the screening visit
13. Subjects who have had severe gastrointestinal disease (active ulcer, etc.), gastrointestinal surgery, or clinically significant abnormal gastric emptying, or those who have chronically used medications that directly affect gastrointestinal motility within 24 weeks prior to the screening visit (However, those with a history of appendectomy or cholecystectomy are eligible to participate)
14. Subjects with a history of acute or chronic pancreatitis (e.g., acute and chronic pancreatitis, symptomatic cholecystitis, pancreatic injury, etc.)
15. Subjects with a history of malignant tumor within the past 5 years

    * Those who have been assessed as having achieved complete remission (CR, pCR) of the tumor and have remained free of recurrence for ≥5 years from the date of assessment are eligible to participate
    * Those with a history of thyroid cancer, excluding medullary thyroid carcinoma (MTC), carcinoma in situ of cervix, or basal cell or squamous cell carcinoma within the past 5 years are eligible to participate
16. Subjects with a history of major depressive disorder, anxiety disorder, or other severe mental illness (e.g., schizophrenia, bipolar disorder, etc.) in an unstable state
17. Subjects who tested positive for HBsAg, HCV antibody, or HIV antibody at the screening visit (However, those who tested positive for HCV-Ab but negative for HCV-RNA may participate.)
18. Subjects whose test results meet the following at the screening visit and pre-randomization testing:

    * Uncontrolled hypertension: siSBP≥160 mmHg or siDBP≥100 mmHg
    * AST or ALT > 3 times the upper limit of normal , total bilirubin > 2 times the upper limit of normal
    * Amylase or Lipase > 3 times the upper limit of normal
    * eGFR ≤ 45mL/min/1.73m²
    * TG > 500 mg/dL (or 5.65 mmol/L)
    * Fasting C-peptide < 0.6 ng/mL (or 0.2 nmol/L)
    * Hemoglobin <11.0 g/dL (male), <10.0 g/dL (female)
    * Calcitonin ≥ 100 ng/L (or 100 pg/mL)
19. Subjects with hematologic conditions (e.g., hemolytic anemia, hemoglobinopathies) that may interfere with HbA1c measurements at the screening visit and pre-randomization testing
20. Subjects with a history of alcoholism or substance abuse
21. Subjects who have taken systemic steroids or growth hormones for 7 days or more (including oral and intravenous administration) within 8 weeks prior to the screening visit
22. Subjects with a history of resistance or hypersensitivity to the drugs in the same class as the investigational product
23. Subjects who have received other investigational products or used investigational devices within 12 weeks prior to the screening visit
24. Subjects who have donated blood, had significant bleeding (>400 mL), or received blood transfusion or blood products within 12 weeks prior to the screening visit
25. Subjects with a history of nonarteritic anterior ischemic optic neuropathy (NAION)
26. Subjects with a positive pregnancy test, pregnant women, or lactating women
27. Subjects who deemed ineligible as subjects by the investigator for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
A change in HbA1c from baseline at Week 24 | Baseline, 24 Weeks

SECONDARY OUTCOMES:
A change in HbA1c from baseline at each time point at Weeks 4, 8, 12, and 16 | Baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks
Proportion of subjects with HbA1c <7% at week 24 | 24 weeks
Proportion of subjects with HbA1c ≤6.5% at week 24 | 24 weeks
A change in glucose metabolism indicators from baseline at week 24 | Baseline, 24 weeks
  FPG, fasting insulin, HOMA-IR, HOMA-β (However, percent changes in fasting insulin, HOMA-IR, and HOMA-β are also presented)
A percent change in lipids from baseline at week 24 | Baseline, 24 weeks
  TG, LDL-C, HDL-C
A change in blood pressure from baseline at week 24 | Baseline, 24 weeks
  sitSBP, sitDBP
A change in body weight from baseline at week 24 | Baseline, 24 weeks
A percent change in body weight from baseline at week 24 | Baseline, 24 weeks
A change in waist circumference from baseline at week 24 | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Rae Kim, Principal Investigator — Bucheon St. Mary Hospital, The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No